CLINICAL TRIAL: NCT07406256
Title: Safety and Efficacy of the AviClear Laser System for the Treatment of Sebaceous Hyperplasia
Brief Title: A Device Study for the Treatment of Sebaceous Hyperplasia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-25-SH02
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Sebaceous Hyperplasia

STUDY DESIGN:
Masking Description: Outcome Assessor is blinded to study design and time point being assessed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Laser Treatment (Experimental)
  Interventions: Device: Cutera Laser System

INTERVENTIONS:
Device: Cutera Laser System — Subjects will receive laser treatments

SUMMARY:
To evaluate the safety and efficacy of the AviClear laser system for the treatment of sebaceous hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects is 18-80 years of age (inclusive) and Fitzpatrick Skin Types I-VI.
2. Subject has a minimum of one clinically diagnosed Sebaceous Hyperplasia lesion and up to ten lesions to be treated on their face, excluding within the orbital rim, scalp, or nose, as determined by the Investigator and/or expert evaluator.
3. Subject is willing to have SH lesion(s) treated and understands that their lesion(s) may undergo additional treatment sessions at the discretion of the Investigator at a subsequent visit.
4. Subject must be able to read, speak, and understand English and sign the Informed Consent Form.
5. Subject is willing and able to adhere to the treatment and follow-up schedule and pre/posttreatment care instructions.
6. Subject is willing to have photographs taken of the target area and agrees to the use of photographs for presentation, educational, or marketing purposes. 7. Subject is willing to have videos taken of the study treatment procedure and agree to the use of videos for presentation, educational, or marketing purposes.

8. Subject agrees to refrain from using all other lesion removal products or treatments (e.g., retinols, retinoids, exfoliating products) to the treated SH lesions or any new SH lesions during the study period.

9. Subject is willing to have very limited sun exposure (including avoiding tanning booths, sun lamps, sunbathing) and use an Investigator approved sunblock or sunscreen of SPF 30 or higher on the treatment area every day for the duration of the study, including the follow-up period.

10. Subject agrees to not undergo any other procedure(s) or add any new treatment modalities in the target area during the study.

Exclusion Criteria:

1. Subject has participated in a clinical trial treating the target area within 1 month prior to study participation.
2. Subject has received injections of botulinum toxin, collagen, hyaluronic acid filler, or dermal fillers in the target area within 1 month prior to study participation.
3. Subject has undergone prior treatments for any reason to the target area within 3 months of study participation, such as deep chemical peels, dermabrasion, microneedling, radiofrequency treatment, laser or light-based procedures, cryodestruction or chemodestruction, intralesional steroids, photodynamic therapy, electrodessication, or surgery.
4. Subject has used topical lesion removal products (e.g., retinols, retinoids, exfoliating products) within 2 weeks of study participation and/or systemic use of retinoid, such as isotretinoin, within 6 months of study participation.
5. Subject was treated previously with AviClear for SH lesions.
6. Subject has history of diagnosed immunosuppression/immune deficiency disorders or currently using prednisone or anti-rejection medications.
7. Subject has history of malignant tumors in the target area.
8. Subject has history of suffering from diagnosed coagulation disorders or taking prescription anticoagulation medications. Low dose (81mg) aspirin is permitted.
9. Subject has history of diagnosed connective tissue disease, such as systemic lupus erythematosus or scleroderma.
10. Subject has personal history or Family History of Muir-Torre Syndrome or with a known history of multiple family members (including parents, grandparents, siblings, or children) with colon cancer at discretion of Investigator.
11. Subject has history of Basal Cell Nevus Syndrome.
12. Subject has history of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the target area, unless treatment is conducted following a prophylactic regimen.
13. Subject has history of radiation to the target area, currently undergoing treatment for skin cancer in the target area or undergoing chemotherapy for the treatment of any cancer.
14. Subject has any use of medication(s) that is known to increase sensitivity to light according to Investigator's discretion.
15. Subject is prone to developing hypertrophic scars or to be keloid producer. 16. Subject has presence of any skin condition in the target area (e.g. eczema, psoriasis, dermatitis, rash, papulo-pustular rosacea, infection, open wounds, irregular or atypical moles, questionable pigmented lesions) that would interfere with the diagnosis or assessment of SH.

17. Subject has excessive hair in the target area (e.g. beards, sideburns, moustaches, scalp, etc.) that would interfere with diagnosis or assessment of SH in the target area (okay if shaved).

18. Subject is excessively tanned on the target area or unable/unlikely to refrain from tanning on the target area during the study.

19. Subject has tattoos or permanent makeup on the target area. 20. Subject has a metal or electronic implant under the skin in the target area. 21. Subject is pregnant and/or breastfeeding or planning to become pregnant during the study.

22. As per the Investigator's discretion, any physical, mental, or medical condition that might make it unsafe for the subject to participate in this study or might interfere with subject's participation in the full study protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
GAIS Response Rate of Treated Lesions | 8-weeks post final treatment
  The primary outcome measure to evaluate the efficacy of the AviClear device is the GAIS response rate of treated SH lesions at 8-weeks post final treatment.